CLINICAL TRIAL: NCT02352363
Title: A Phase 3, Randomized Study Investigating the Safety of CVT-301 (Levodopa Inhalation Powder) in Parkinson's Disease (PD) Patients With Motor Response Fluctuations (OFF Phenomena) Compared to an Observational Cohort Control
Brief Title: Randomized Safety Study of CVT-301 Compared to an Observational Control Group
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVT-301-005
Record Dates: First submitted 2015-01-26; First posted 2015-02-02 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's Disease; Motor fluctuations; levodopa; inhaled drugs; OFF episodes
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CVT-301 (Experimental): Capsules of Levodopa Inhalational Powder (LIP) used up to 5 times per day for OFF episodes, for up to 54 weeks duration.
  Interventions: Drug: CVT-301
- Observational Cohort (Other): Standard of care. Patients in both the CVT-301 treatment group and the observational cohort will be managed with their standard PD treatment throughout the study.
  Interventions: Other: Observational cohort

INTERVENTIONS:
Drug: CVT-301
  Other Names: Inhaled levodopa
  Arms: CVT-301
Other: Observational cohort
  Arms: Observational Cohort

SUMMARY:
This study is a 12-month, open-label, randomized, multicenter study which will evaluate the safety and efficacy of CVT-301 for the treatment of up to 5 OFF episodes per day in Parkinson's Disease (PD) patients experiencing motor fluctuations (OFF episodes) and will include a concurrent observational cohort of PD patients managed using the usual standards of care.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, Phase 2b study in patients with PD (CVT-301-003) demonstrated clinically important, and statistically significant CVT-301-associated improvements in motor function at doses of 35 and 50 mg LD FPD, compared with placebo, as measured by the Unified Parkinson's Disease Rating Scale (UPDRS) motor assessment (Part 3); furthermore, CVT-301 was generally safe and well tolerated. A Phase 3, randomized, placebo-controlled study designed to assess the efficacy and safety of 35 mg and 50 mg FPD as an adjunct to a CD/LD regimen in the treatment of OFF symptoms over 12 weeks (CVT-301-004) was conducted in parallel with this study.

ELIGIBILITY:
Inclusion Criteria:

* Has signed and dated an Internal Review Board/Independent Ethics Committee (IRB/IEC)-approved informed consent form before any protocol-specific screening procedures are performed.
* Women of child-bearing potential must use protocol-defined contraceptive measures and must have a negative serum human chorionic gonadotropin (hCG) test at screening. These patients must be willing to remain on their current form of contraception for the duration of the study.
* Patients who have idiopathic PD (i.e., not induced by drugs or other diseases) as defined by fulfilling Steps 1 and 2 of the United Kingdom (UK) Brain Bank criteria, diagnosed after the age of 30 years.
* Patients who are classified as Stage 1 to 3 (in the ON state) on the modified Hoehn and Yahr scale for staging of PD severity.
* Patients who have experienced motor fluctuations for a minimum of 2 hours of average daily OFF time per waking day (excluding early morning OFF time) by self-report and confirmed by the PD Diary (on 3 consecutive days) during the screening period.

Exclusion Criteria:

* Patients who have dyskinesia of a severity that would significantly interfere with their ability to participate or perform study procedures.
* Pregnant or lactating females or females wishing to become pregnant.
* Patients who have any known contraindication to the use of levodopa (LD), including a history of malignant melanoma or a history of narrow-angle glaucoma.
* Patients who have had previous surgery for PD (including but not limited to deep brain stimulation [DBS] or cell transplantation).
* Patients with a history of psychotic symptoms requiring treatment, or suicide ideation or attempt within the prior 12 months.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Oh, MD, Study Director — Acorda Therapeutics
Locations (76):
- United States (14):
  - Acorda Site #7145, Scottsdale, Arizona
  - Acorda Site # 7142, Fountain Valley, California
  - Acorda Site #7139, Panorama City, California
  - Acorda Site #7141, Sunnyvale, California
  - Acorda Site #7137, Ormond Beach, Florida
  - Acorda Site #7135, St. Petersburg, Florida
  - Acorda Site #7130, Sunrise, Florida
  - Acorda Site #7133, Atlanta, Georgia
  - Acorda Site #7134, Atlanta, Georgia
  - Acorda Site #7131, Decatur, Georgia
  - Acorda Site #7138, Honolulu, Hawaii
  - Acorda Site #7140, Des Moines, Iowa
  - Acorda Site #7150, Baton Rouge, Louisiana
  - Acorda Site #7148, Toledo, Ohio
- Austria (3):
  - Acorda Site #7004, Innsbruck
  - Acorda Site #7002, Linz
  - Acorda Site #7003, Vienna
- Belgium (3):
  - Acorda Site #7011, Brussels
  - Acorda Site #7012, Edegem
  - Acorda Site #7013, Ghent
- Czechia (5):
  - Acorda Site #7024, Choceň
  - Acorda Site #7025, Ostrava
  - Acorda Site #7021, Pardubice
  - Acorda Site #7022, Prague
  - Acorda Site #7023, Rychnov nad Kněžnou
- France (7):
  - Acorda Site #7036, Amiens
  - Acorda Site #7037, Bordeaux
  - Acorda Site #7034, Marseille
  - Acorda Site #7031, Montpellier
  - Acorda Site #7033, Nîmes
  - Acorda Site #7032, Strasbourg
  - Acorda Site #7035, Toulouse
- Germany (9):
  - Acorda Site #7041, Achim
  - Acorda Site #7043, Beelitz-Heilstätten
  - Acorda Site #7049, Berlin
  - Acorda Site #7050, Bochum
  - Acorda Site #7048, Bremerhaven
  - Acorda Site #7047, Cologne
  - Acorda Site #7046, Marburg
  - Acorda Site #7042, Munich
  - Acorda Site #7044, Ulm
- Hungary (2):
  - Acorda Site #7053, Budapest
  - Acorda Site #7051, Budapest
- Israel (4):
  - Acorda Site #7062, Jerusalem
  - Acorda Site #7064, Petah Tikva
  - Acorda Site #7061, Ramat Gan
  - Acorda Site #7063, Tel Aviv
- Acorda Site #7045, The Hague, Netherlands
- Poland (8):
  - Acorda Site #7085, Gdansk
  - Acorda Site #7084, Katowice
  - Acorda Site #7083, Kracow
  - Acorda Site #7086, Krakow
  - Acorda Site #7087, Krakow
  - Acorda Site #7082, Lodz
  - Acorda Site #7081, Warsaw
  - Acorda Site #7088, Warsaw
- Romania (5):
  - Acorda Site #7094, Brasov
  - Acorda Site #7092, Brasov
  - Acorda Site #7093, Bucharest
  - Acorda Site #7091, Constanța
  - Acorda Site #7095, Târgu Mureş
- Serbia (3):
  - Acorda Site #7101, Belgrade
  - Acorda Site #7102, Belgrade
  - Acorda Site #7103, Kragujevac
- Spain (9):
  - Acorda Site #7112, Sant Cugat del Vallès, Barcelona
  - Acorda Site #7116, Barcelona
  - Acorda Site #7111, Barcelona
  - Acorda Site #7120, Barcelona
  - Acorda Site #7119, Barcelona
  - Acorda Site #7113, Burgos
  - Acorda Site #7115, Donostia / San Sebastian
  - Acorda Site #7118, Madrid
  - Acorda Site #7114, Madrid
- United Kingdom (3):
  - Acorda Site #7123, Cambridge
  - Acorda Site #7121, Glasgow
  - Acorda Site #7122, London

REFERENCES:
- [Derived] Kaminsky DA, Grosset DG, Kegler-Ebo DM, Cangiamilla S, Klingler M, Zhao P, Oh C. Natural history of lung function over one year in patients with Parkinson's disease. Respir Med. 2021 Jun;182:106396. doi: 10.1016/j.rmed.2021.106396. Epub 2021 Apr 16. PMID 33866196
- See also: Click here for more information about this study:CVT-301-005 — http://cvt301.acordatrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 408 of the 513 screened were randomly assigned to CVT-301 (278) or observational cohort (130). Of these 408 patients, 398 received at least 1 dose of inhaled CVT-301 CVT-treatment group) or came in for OV1 (observational cohort) and were included in the Safety Population.
Groups:
- CVT-301: Capsules of Levodopa Inhalational Powder (LIP) used up to 5 times per day for OFF episodes, for up to 54 weeks duration.
  CVT-301
- Observational Cohort: Standard of care. Patients in both the CVT-301 treatment group and the observational cohort will be managed with their standard PD treatment throughout the study.
  Observational cohort
Period: Overall Study
Arm/Group | CVT-301 | Observational Cohort
Started | 278 | 130
Completed | 271 | 127
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Population: A total of 408 of the 513 screened were randomly assigned to CVT-301 (278) or observtional cohort (130). Of these 408 patients, 398 received at least 1 dose of inhaled CVT-301 (CVT-treatment group) or came in for OV1 (observational cohort) and were included in the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVT-301 | Observational Cohort | Total
Number analyzed (Participants) | 271 | 127 | 398
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 137 | 59 | 196
  >=65 years | 134 | 68 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.54) | 64.2 (7.88) | 63.8 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 49 | 159
  Male | 161 | 78 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 267 | 124 | 391
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 55 | 34 | 89
  Hungary | 5 | 0 | 5
  Czechia | 22 | 16 | 38
  United States | 21 | 6 | 27
  United Kingdom | 4 | 5 | 9
  Spain | 28 | 8 | 36
  Austria | 11 | 1 | 12
  Belgium | 4 | 1 | 5
  Poland | 61 | 32 | 93
  Israel | 15 | 6 | 21
  France | 13 | 7 | 20
  Serbia | 11 | 4 | 15
  Germany | 21 | 7 | 28
Spirometry FEV1 [Mean (Standard Deviation); unit: Liters] | 2.842 (0.7538) | 2.838 (0.853) | 2.841 (0.7831)
Spirometry FVC [Mean (Standard Deviation); unit: Liters] | 3.665 (0.9203) | 3.696 (1.0497) | 3.675 (0.9622)
Spirometry FEV1/FVC [Mean (Standard Deviation); unit: Ratio %] | 77.6 (6.23) | 76.8 (6.50) | 77.3 (6.32)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Safety Assessed by Forced Expiratory Volume in 1 Second [FEV1]
Description: To characterize the pulmonary safety, as assessed by spirometry (forced expiratory volume in 1 second [FEV1], over a 12 month period.
Time Frame: Month 12 reported
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CVT-301 | Observational Cohort
Number analyzed (Participants) | 271 | 127
Liters | 2.778 (0.7309) | 2.767 (0.8419)

2. Primary Outcome: Pulmonary Safety Assessed by Forced Vital Capacity [FVC].
Description: To characterize the pulmonary safety, as assessed by spirometry (forced vital capacity).
Time Frame: Month 12 reported
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CVT-301 | Observational Cohort
Number analyzed (Participants) | 271 | 127
Liters | 3.558 (0.8987) | 3.642 (1.0687)

3. Primary Outcome: Pulmonary Safety Assessed by Forced Expiratory Volume in 1 Second / Forced Vital Capacity Ratio.
Description: To characterize the pulmonary safety, as assessed by spirometry (forced expiratory volume in 1 second / forced vital capacity ratio).
Time Frame: Month 12 reported
Measure: Mean (Standard Deviation); unit: Ratio (%)
Arm/Group | CVT-301 | Observational Cohort
Number analyzed (Participants) | 271 | 127
Ratio (%) | 78.1 (6.04) | 76.1 (6.4)

4. Secondary Outcome: Diffusion Capacity of the Lungs for Carbon Monoxide (DLco).
Description: To describe the effects of CVT-301 on diffusion capacity of the lungs for carbon monoxide (DLco) over a 12-month period.
Time Frame: Month 12 reported
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | CVT-301 | Observational Cohort
Number analyzed (Participants) | 271 | 127
mL/min/mmHg | 23.273 (6.0025) | 23.473 (7.0848)

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | CVT-301 | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 1/271 | 0/127
Serious Adverse Events (participants affected / at risk) | 42/271 | 13/127
Other Adverse Events (participants affected / at risk) | 192/271 | 64/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVT-301 (N=271) | Observational Cohort (N=127)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Parkinson's disease (Nervous system disorders) | 2 (2) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedure haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Astenia (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVT-301 (N=271) | Observational Cohort (N=127)
Nasopharyngitis (Infections and infestations) | 18 (20) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 13 (16) | 3 (3)
Bronchitis (Infections and infestations) | 7 (7) | 4 (6)
Influenza (Infections and infestations) | 4 (5) | 4 (4)
Dyskinesia (Nervous system disorders) | 17 (18) | 5 (5)
Parkinson's disease (Nervous system disorders) | 8 (8) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (19) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (43) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 22 (28) | 7 (8)
Nausea (Gastrointestinal disorders) | 10 (12) | 1 (1)
Hypertension (Vascular disorders) | 9 (9) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 7 (12) | 4 (4)
Blood pressure increased (Investigations) | 1 (1) | 4 (5)
Vertigo (Ear and labyrinth disorders) | 8 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT02352363/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT02352363/SAP_001.pdf